CLINICAL TRIAL: NCT00005136
Title: Family Heart Study (FHS)
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1006; U01HL056564 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Coronary Disease; Heart Diseases

SUMMARY:
To identify and evaluate genetic and non-genetic determinants of coronary heart disease (CHD), atherosclerosis, and their risk factors in ongoing population-based epidemiology studies. The multicenter study was conducted in three phases which were: Phase I, the family history component: Phase II, the clinical examination and follow-up component; and Phase III, the molecular genetic and genetic epidemiology studies component.

DETAILED DESCRIPTION:
BACKGROUND:

Advances in molecular genetics, genetic epidemiology, population genetics, and identification of new risk factors and clusters of risk factors for cardiovascular disease made 1991 an opportune time to take advantage of the extensive information about cardiovascular disease, pre-clinical atherosclerosis, and risk factors in individuals who had been examined in ongoing, state-of-the-art epidemiological studies supported by the NHLBI. By recruiting first degree relatives of random samples of such defined populations, FHS obtained information about familial aggregation, genetic and environmental contributions to variance in continuous variables, and the frequency and distribution of elevated levels of risk factors and of selected major genes in the general population.

The FHS was initiated by staff and approved by the Clinical Applications and Prevention Advisory Commitee in May, 1990. The Requests for Proposals were released in July 1991. Contracts were awarded in June, 1992.

DESIGN NARRATIVE:

During Phases I and II from May 1992-May 1996, probands, aged 45-69, were recruited from the Framingham Heart Study, the Utah Family Tree Study and the North Carolina and Minnesota sites of the ARIC Study, along with their relatives, for participation in the Family Heart Study. Two groups of probands were selected, either randomly or by a high family risk of CHD as calculated from data from the parent study. Additional family structure and disease history data were collected on 3,150 probands and 22,909 of their relatives. Clinical examination and follow-up of these random and high CHD risk families were conducted on a total of 1,253 families including 5,975 individuals, of whom 102 families including 265 individuals were African-American. The examinations included information on anthropometry, blood pressure, ECG, carotid ultrasound, pulmonary function, and blood chemistries. Questionnaire data included medical and reproductive histories, diet, physical activity, tobacco and alcohol consumption, education, income and psychosocial factors including hostility, social support and stress. Phases I and II included four field centers, a coordinating center, and a central blood laboratory.

In August 1996, Phase III began when cooperative agreements were awarded to a consortium of seven investigator-initiated grants to conduct molecular genetic and genetic epidemiology studies using data collected during Phases I and II. Phase III ended in July 2001. The objective of Phase III was to perform molecular genetic and genetic epidemiology studies using the extensive data on family and medical histories, risk factors, life style, blood specimens, and banked DNA previously collected by the FHS. Studies included novel molecular genetics of candidate genes and genome-wide searches with anonymous markers for the detection, mapping, and characterization of coronary heart disease and atherosclerosis genes. Genetic epidemiology analyses were conducted that contributed new information on the familial aspects of atherosclerosis and intermediate phenotypes in African Americans. Phase III also included four field centers, a central laboratory, a molecular genetics laboratory, and a coordinating center.

The study was renewed in 2001 as the Family Heart Study - Subclinical Atherosclerosis Network (FHS-SCAN) to complete analyses of genome-wide scan data and to genotype promising markers. The study expects to enroll 401 informative pedigrees (3,027 individuals) previously examined and genotyped by the NHLBI Family Heart Study to quantify coronary and aortic calcium volume in order to identify genes associated with atherosclerosis. In addition, 315 African American sibships (770 individuals) previously examined and comparably genotyped by the Hypertension Epidemiology Network (HyperGEN) will be examined at one study center to address these study questions in this minority population.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-06; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Arnett — University of Minnesota; John Eckfeldt — University of Minnesota; R. Ellison — Boston University; Aaron Folsom — University of Minnesota; Gerardo Heiss — University of North Carolina; Steven Hunt — University of Utah; Mark Leppert — University of Utah; Michael Province — Washington University School of Medicine; D.C. Rao — Washington University School of Medicine; Roger Williams — University of Utah

REFERENCES:
- [Background] Jacques PF, Bostom AG, Williams RR, Ellison RC, Eckfeldt JH, Rosenberg IH, Selhub J, Rozen R. Relation between folate status, a common mutation in methylenetetrahydrofolate reductase, and plasma homocysteine concentrations. Circulation. 1996 Jan 1;93(1):7-9. doi: 10.1161/01.cir.93.1.7. PMID 8616944
- [Background] Pankow JS, Folsom AR, Province MA, Rao DC, Eckfeldt J, Heiss G, Shahar E, Wu KK. Family history of coronary heart disease and hemostatic variables in middle-aged adults. Atherosclerosis Risk in Communities Investigators and Family Heart Study Research Group. Thromb Haemost. 1997 Jan;77(1):87-93. PMID 9031455
- [Background] Higgins M, Province M, Heiss G, Eckfeldt J, Ellison RC, Folsom AR, Rao DC, Sprafka JM, Williams R. NHLBI Family Heart Study: objectives and design. Am J Epidemiol. 1996 Jun 15;143(12):1219-28. doi: 10.1093/oxfordjournals.aje.a008709. PMID 8651220
- [Background] Borecki IB, Province MA, Rao DC. Power of segregation analysis for detection of major gene effects on quantitative traits. Genet Epidemiol. 1994;11(5):409-18. doi: 10.1002/gepi.1370110503. PMID 7835687
- [Background] Borecki IB, Province MA, Rao DC. Inferring a major gene for quantitative traits by using segregation analysis with tests on transmission probabilities: how often do we miss? Am J Hum Genet. 1995 Jan;56(1):319-26. PMID 7825593
- [Background] Wilk JB, Djousse L, Borecki I, Atwood LD, Hunt SC, Rich SS, Eckfeldt JH, Arnett DK, Rao DC, Myers RH. Segregation analysis of serum uric acid in the NHLBI Family Heart Study. Hum Genet. 2000 Mar;106(3):355-9. doi: 10.1007/s004390000243. PMID 10798367
- [Background] Kronenberg F, Rich SS, Sholinsky P, Arnett DK, Province ME, Myers RH, Eckfeldt JH, Williams RR, Hunt SC. Insulin and hypertension in the NHLBI Family Heart Study: a sibpair approach to a controversial issue. Am J Hypertens. 2000 Mar;13(3):240-50. doi: 10.1016/s0895-7061(99)00177-6. PMID 10777027
- [Background] Weidner G, Rice T, Knox SS, Ellison RC, Province MA, Rao DC, Higgins MW. Familial resemblance for hostility: the National Heart, Lung, and Blood Institute Family Heart Study. Psychosom Med. 2000 Mar-Apr;62(2):197-204. doi: 10.1097/00006842-200003000-00008. PMID 10772397
- [Background] Coon H, Leppert MF, Kronenberg F, Province MA, Myers RH, Arnett DK, Eckfeldt JH, Heiss G, Williams RR, Hunt SC. Evidence for a major gene accounting for mild elevation in LDL cholesterol: the NHLBI Family Heart Study. Ann Hum Genet. 1999 Sep;63(Pt 5):401-12. doi: 10.1046/j.1469-1809.1999.6350401.x. PMID 10735582
- [Background] Hong Y, Leppert MF, Lin J, Hunt SC, Rich SS, Arnett DK, Myers RH, Eckfeldt J, Williams RR, Province MA. No evidence of linkage between the very-low-density lipoprotein receptor gene and fasting serum insulin or homeostasis model assessment insulin resistance index: the National Heart, Lung, and Blood Institute Family Heart Study. Metabolism. 2000 Mar;49(3):293-7. doi: 10.1016/s0026-0495(00)90022-2. PMID 10726903
- [Background] Li R, Bensen JT, Hutchinson RG, Province MA, Hertz-Picciotto I, Sprafka JM, Tyroler HA. Family risk score of coronary heart disease (CHD) as a predictor of CHD: the Atherosclerosis Risk in Communities (ARIC) study and the NHLBI family heart study. Genet Epidemiol. 2000 Mar;18(3):236-50. doi: 10.1002/(SICI)1098-2272(200003)18:33.0.CO;2-0. PMID 10723108
- [Background] Ellison RC, Myers RH, Zhang Y, Djousse L, Knox S, Williams RR, Province MA. Effects of similarities in lifestyle habits on familial aggregation of high density lipoprotein and low density lipoprotein cholesterol: the NHLBI Family Heart Study. Am J Epidemiol. 1999 Nov 1;150(9):910-8. doi: 10.1093/oxfordjournals.aje.a010099. PMID 10547136
- [Background] Bensen JT, Liese AD, Rushing JT, Province M, Folsom AR, Rich SS, Higgins M. Accuracy of proband reported family history: the NHLBI Family Heart Study (FHS). Genet Epidemiol. 1999;17(2):141-50. doi: 10.1002/(SICI)1098-2272(1999)17:23.0.CO;2-Q. PMID 10414557
- [Background] Siegmund KD, Todorov AA, Province MA. A frailty approach for modelling diseases with variable age of onset in families: the NHLBI Family Heart Study. Stat Med. 1999 Jun 30;18(12):1517-28. doi: 10.1002/(sici)1097-0258(19990630)18:123.0.co;2-4. PMID 10398289
- [Background] Ellison RC, Zhang Y, Myers RH, Swanson JL, Higgins M, Eckfeldt J. Lewis blood group phenotype as an independent risk factor for coronary heart disease (the NHLBI Family Heart Study). Am J Cardiol. 1999 Feb 1;83(3):345-8. doi: 10.1016/s0002-9149(98)00866-2. PMID 10072221
- [Background] Hopkins PN, Hunt SC, Schreiner PJ, Eckfeldt JH, Borecki IB, Ellison CR, Williams RR, Siegmund KD. Lipoprotein(a) interactions with lipid and non-lipid risk factors in patients with early onset coronary artery disease: results from the NHLBI Family Heart Study. Atherosclerosis. 1998 Dec;141(2):333-45. doi: 10.1016/s0021-9150(98)00174-9. PMID 9862182
- [Background] Knox SS, Siegmund KD, Weidner G, Ellison RC, Adelman A, Paton C. Hostility, social support, and coronary heart disease in the National Heart, Lung, and Blood Institute Family Heart Study. Am J Cardiol. 1998 Nov 15;82(10):1192-6. doi: 10.1016/s0002-9149(98)00599-2. PMID 9832093
- [Background] Pankow JS, Folsom AR, Province MA, Rao DC, Williams RR, Eckfeldt J, Sellers TA. Segregation analysis of plasminogen activator inhibitor-1 and fibrinogen levels in the NHLBI family heart study. Arterioscler Thromb Vasc Biol. 1998 Oct;18(10):1559-67. doi: 10.1161/01.atv.18.10.1559. PMID 9763527
- [Background] Djousse L, Ellison RC, Zhang Y, Arnett DK, Sholinsky P, Borecki I. Relation between dietary fiber consumption and fibrinogen and plasminogen activator inhibitor type 1: The National Heart, Lung, and Blood Institute Family Heart Study. Am J Clin Nutr. 1998 Sep;68(3):568-75. doi: 10.1093/ajcn/68.3.568. PMID 9734732
- [Background] Garg UC, Arnett DK, Evans G, Eckfeldt JH. No association between factor V Leiden mutation and coronary heart disease or carotid intima media thickness: the NHLBI Family Heart Study. Thromb Res. 1998 Mar 15;89(6):289-93. doi: 10.1016/s0049-3848(98)00019-x. No abstract available. PMID 9669751
- [Background] Folsom AR, Pankow JS, Williams RR, Evans GW, Province MA, Eckfeldt JH. Fibrinogen, plasminogen activator inhibitor-1, and carotid intima-media wall thickness in the NHLBI Family Heart Study. Thromb Haemost. 1998 Feb;79(2):400-4. PMID 9493598
- [Background] Liao D, Myers R, Hunt S, Shahar E, Paton C, Burke G, Province M, Heiss G. Familial history of stroke and stroke risk. The Family Heart Study. Stroke. 1997 Oct;28(10):1908-12. doi: 10.1161/01.str.28.10.1908. PMID 9341694
- [Background] Djousse L, Pankow JS, Arnett DK, Zhang Y, Hong Y, Province MA, Ellison RC. Alcohol consumption and plasminogen activator inhibitor type 1: the National Heart, Lung, and Blood Institute Family Heart Study. Am Heart J. 2000 Apr;139(4):704-9. doi: 10.1016/s0002-8703(00)90052-8. PMID 10740155
- [Background] Hunt KJ, Heiss G, Sholinsky PD, Province MA. Familial history of metabolic disorders and the multiple metabolic syndrome: the NHLBI family heart study. Genet Epidemiol. 2000 Dec;19(4):395-409. doi: 10.1002/1098-2272(200012)19:43.0.CO;2-3. PMID 11108648
- [Background] Knox SS, Adelman A, Ellison RC, Arnett DK, Siegmund K, Weidner G, Province MA. Hostility, social support, and carotid artery atherosclerosis in the National Heart, Lung, and Blood Institute Family Heart Study. Am J Cardiol. 2000 Nov 15;86(10):1086-9. doi: 10.1016/s0002-9149(00)01164-4. PMID 11074204
- [Background] Coon H, Myers RH, Borecki IB, Arnett DK, Hunt SC, Province MA, Djousse L, Leppert MF. Replication of linkage of familial combined hyperlipidemia to chromosome 1q with additional heterogeneous effect of apolipoprotein A-I/C-III/A-IV locus. The NHLBI Family Heart Study. Arterioscler Thromb Vasc Biol. 2000 Oct;20(10):2275-80. doi: 10.1161/01.atv.20.10.2275. PMID 11031215
- [Background] Pankow JS, Arnett DK, Borecki IB, Hunt SC, Eckfeldt JH, Folsom AR, Djousse L. Lack of association between the angiotensin-converting enzyme insertion/deletion polymorphism and plasminogen activator inhibitor-1 antigen levels in the National Heart, Lung, and Blood Institute Family Heart Study. Blood Coagul Fibrinolysis. 2000 Sep;11(6):551-8. doi: 10.1097/00001721-200009000-00007. PMID 10997795
- [Background] Djousse L, Myers RH, Coon H, Arnett DK, Province MA, Ellison RC. Smoking influences the association between apolipoprotein E and lipids: the National Heart, Lung, and Blood Institute Family Heart Study. Lipids. 2000 Aug;35(8):827-31. doi: 10.1007/s11745-000-0591-1. PMID 10984105
- [Background] Feitosa MF, Borecki I, Hunt SC, Arnett DK, Rao DC, Province M. Inheritance of the waist-to-hip ratio in the National Heart, Lung, and Blood Institute Family Heart Study. Obes Res. 2000 Jul;8(4):294-301. doi: 10.1038/oby.2000.35. PMID 10933305
- [Background] Tsai MY, Arnett DK, Eckfeldt JH, Williams RR, Ellison RC. Plasma homocysteine and its association with carotid intimal-medial wall thickness and prevalent coronary heart disease: NHLBI Family Heart Study. Atherosclerosis. 2000 Aug;151(2):519-24. doi: 10.1016/s0021-9150(99)00409-8. PMID 10924729
- [Background] Salomaa V, Pankow J, Heiss G, Cakir B, Eckfeldt JH, Ellison RC, Myers RH, Hiller KM, Brantley KR, Morris TL, Weston BW. Genetic background of Lewis negative blood group phenotype and its association with atherosclerotic disease in the NHLBI family heart study. J Intern Med. 2000 Jun;247(6):689-98. doi: 10.1046/j.1365-2796.2000.00682.x. PMID 10886491
- [Background] Wilk JB, Djousse L, Arnett DK, Rich SS, Province MA, Hunt SC, Crapo RO, Higgins M, Myers RH. Evidence for major genes influencing pulmonary function in the NHLBI family heart study. Genet Epidemiol. 2000 Jul;19(1):81-94. doi: 10.1002/1098-2272(200007)19:13.0.CO;2-8. PMID 10861898
- [Background] Hong Y, Rautaharju PM, Hopkins PN, Arnett DK, Djousse L, Pankow JS, Sholinsky P, Rao DC, Province MA. Familial aggregation of QT-interval variability in a general population: results from the NHLBI Family Heart Study. Clin Genet. 2001 Mar;59(3):171-7. doi: 10.1034/j.1399-0004.2001.590305.x. PMID 11260226
- [Background] Hunt SC, Kronenberg F, Eckfeldt JH, Hopkins PN, Myers RH, Heiss G. Association of plasma bilirubin with coronary heart disease and segregation of bilirubin as a major gene trait: the NHLBI family heart study. Atherosclerosis. 2001 Feb 15;154(3):747-54. doi: 10.1016/s0021-9150(00)00420-2. PMID 11257278
- [Background] Pankow JS, Folsom AR, Cushman M, Borecki IB, Hopkins PN, Eckfeldt JH, Tracy RP. Familial and genetic determinants of systemic markers of inflammation: the NHLBI family heart study. Atherosclerosis. 2001 Feb 15;154(3):681-9. doi: 10.1016/s0021-9150(00)00586-4. PMID 11257270
- [Background] Peacock JM, Arnett DK, Atwood LD, Myers RH, Coon H, Rich SS, Province MA, Heiss G. Genome scan for quantitative trait loci linked to high-density lipoprotein cholesterol: The NHLBI Family Heart Study. Arterioscler Thromb Vasc Biol. 2001 Nov;21(11):1823-8. doi: 10.1161/hq1101.097804. PMID 11701472
- [Background] Feitosa MF, Borecki IB, Rich SS, Arnett DK, Sholinsky P, Myers RH, Leppert M, Province MA. Quantitative-trait loci influencing body-mass index reside on chromosomes 7 and 13: the National Heart, Lung, and Blood Institute Family Heart Study. Am J Hum Genet. 2002 Jan;70(1):72-82. doi: 10.1086/338144. Epub 2001 Nov 16. PMID 11713718
- [Background] Folsom AR, Pankow JS, Tracy RP, Arnett DK, Peacock JM, Hong Y, Djousse L, Eckfeldt JH; Investigators of the NHBLI Family Heart Study. Association of C-reactive protein with markers of prevalent atherosclerotic disease. Am J Cardiol. 2001 Jul 15;88(2):112-7. doi: 10.1016/s0002-9149(01)01603-4. PMID 11448405
- [Background] Kronenberg F, Pereira MA, Schmitz MK, Arnett DK, Evenson KR, Crapo RO, Jensen RL, Burke GL, Sholinsky P, Ellison RC, Hunt SC. Influence of leisure time physical activity and television watching on atherosclerosis risk factors in the NHLBI Family Heart Study. Atherosclerosis. 2000 Dec;153(2):433-43. doi: 10.1016/s0021-9150(00)00426-3. PMID 11164433
- [Background] Djousse L, Myers RH, Province MA, Hunt SC, Eckfeldt JH, Evans G, Peacock JM, Ellison RC. Influence of apolipoprotein E, smoking, and alcohol intake on carotid atherosclerosis: National Heart, Lung, and Blood Institute Family Heart Study. Stroke. 2002 May;33(5):1357-61. doi: 10.1161/01.str.0000014325.54063.1a. PMID 11988615
- [Background] Djousse L, Pankow JS, Eckfeldt JH, Folsom AR, Hopkins PN, Province MA, Hong Y, Ellison RC. Relation between dietary linolenic acid and coronary artery disease in the National Heart, Lung, and Blood Institute Family Heart Study. Am J Clin Nutr. 2001 Nov;74(5):612-9. doi: 10.1093/ajcn/74.5.612. PMID 11684529
- [Background] Hunt SC, Ellison RC, Atwood LD, Pankow JS, Province MA, Leppert MF. Genome scans for blood pressure and hypertension: the National Heart, Lung, and Blood Institute Family Heart Study. Hypertension. 2002 Jul;40(1):1-6. doi: 10.1161/01.hyp.0000022660.28915.b1. PMID 12105129
- [Background] Kronenberg F, Coon H, Ellison RC, Borecki I, Arnett DK, Province MA, Eckfeldt JH, Hopkins PN, Hunt SC. Segregation analysis of HDL cholesterol in the NHLBI Family Heart Study and in Utah pedigrees. Eur J Hum Genet. 2002 Jun;10(6):367-74. doi: 10.1038/sj.ejhg.5200818. PMID 12080388
- [Background] Coon H, Eckfeldt JH, Leppert MF, Myers RH, Arnett DK, Heiss G, Province MA, Hunt SC. A genome-wide screen reveals evidence for a locus on chromosome 11 influencing variation in LDL cholesterol in the NHLBI Family Heart Study. Hum Genet. 2002 Sep;111(3):263-9. doi: 10.1007/s00439-002-0773-8. Epub 2002 Jul 31. PMID 12215839
- [Background] Djousse L, Rothman KJ, Cupples LA, Arnett DK, Ellison RC; NHLBI Family Heart Study. Relation between serum albumin and carotid atherosclerosis: the NHLBI Family Heart Study. Stroke. 2003 Jan;34(1):53-7. doi: 10.1161/01.str.0000048675.97975.84. PMID 12511750
- [Background] Jacques PF, Bostom AG, Selhub J, Rich S, Ellison RC, Eckfeldt JH, Gravel RA, Rozen R; National Heart, Lung and Blood Institute, National Institutes of Health. Effects of polymorphisms of methionine synthase and methionine synthase reductase on total plasma homocysteine in the NHLBI Family Heart Study. Atherosclerosis. 2003 Jan;166(1):49-55. doi: 10.1016/s0021-9150(02)00204-6. PMID 12482550
- [Background] Djousse L, Folsom AR, Province MA, Hunt SC, Ellison RC; National Heart, Lung, and Blood Institute Family Heart Study. Dietary linolenic acid and carotid atherosclerosis: the National Heart, Lung, and Blood Institute Family Heart Study. Am J Clin Nutr. 2003 Apr;77(4):819-25. doi: 10.1093/ajcn/77.4.819. PMID 12663278
- [Background] Wilk JB, DeStefano AL, Arnett DK, Rich SS, Djousse L, Crapo RO, Leppert MF, Province MA, Cupples LA, Gottlieb DJ, Myers RH. A genome-wide scan of pulmonary function measures in the National Heart, Lung, and Blood Institute Family Heart Study. Am J Respir Crit Care Med. 2003 Jun 1;167(11):1528-33. doi: 10.1164/rccm.200207-755OC. Epub 2003 Mar 13. PMID 12637344
- [Background] Hopkins PN, Heiss G, Ellison RC, Province MA, Pankow JS, Eckfeldt JH, Hunt SC. Coronary artery disease risk in familial combined hyperlipidemia and familial hypertriglyceridemia: a case-control comparison from the National Heart, Lung, and Blood Institute Family Heart Study. Circulation. 2003 Aug 5;108(5):519-23. doi: 10.1161/01.CIR.0000081777.17879.85. Epub 2003 Jul 7. PMID 12847072
- [Background] Djousse L, Arnett DK, Coon H, Province MA, Moore LL, Ellison RC. Fruit and vegetable consumption and LDL cholesterol: the National Heart, Lung, and Blood Institute Family Heart Study. Am J Clin Nutr. 2004 Feb;79(2):213-7. doi: 10.1093/ajcn/79.2.213. PMID 14749225
- [Background] Djousse L, Hunt SC, Arnett DK, Province MA, Eckfeldt JH, Ellison RC. Dietary linolenic acid is inversely associated with plasma triacylglycerol: the National Heart, Lung, and Blood Institute Family Heart Study. Am J Clin Nutr. 2003 Dec;78(6):1098-102. doi: 10.1093/ajcn/78.6.1098. PMID 14668270
- [Background] Knox SS, Wilk JB, Zhang Y, Weidner G, Ellison RC. A genome scan for hostility: the national heart, lung, and blood institute family heart study. Mol Psychiatry. 2004 Feb;9(2):124-6. doi: 10.1038/sj.mp.4001447. No abstract available. PMID 14610523
- [Background] Tang W, Miller MB, Rich SS, North KE, Pankow JS, Borecki IB, Myers RH, Hopkins PN, Leppert M, Arnett DK; National Heart, Lung, and Blood Institute Family Heart Study. Linkage analysis of a composite factor for the multiple metabolic syndrome: the National Heart, Lung, and Blood Institute Family Heart Study. Diabetes. 2003 Nov;52(11):2840-7. doi: 10.2337/diabetes.52.11.2840. PMID 14578304
- [Background] Ellison RC, Zhang Y, Qureshi MM, Knox S, Arnett DK, Province MA; Investigators of the NHLBI Family Heart Study. Lifestyle determinants of high-density lipoprotein cholesterol: the National Heart, Lung, and Blood Institute Family Heart Study. Am Heart J. 2004 Mar;147(3):529-35. doi: 10.1016/j.ahj.2003.10.033. PMID 14999205
- [Background] Coon H, Singh N, Dunn D, Eckfeldt JH, Province MA, Hopkins PN, Weiss R, Hunt SC, Leppert MF; NHLBI Family Heart Study. TXNIP gene not associated with familial combined hyperlipidemia in the NHLBI Family Heart Study. Atherosclerosis. 2004 Jun;174(2):357-62. doi: 10.1016/j.atherosclerosis.2004.02.004. PMID 15136067
- [Background] Pankow JS, Heiss G, Evans GW, Sholinsky P, Province MA, Coon H, Ellison RC, Miller MB, Qaqish B. Familial aggregation and genome-wide linkage analysis of carotid artery plaque: the NHLBI family heart study. Hum Hered. 2004;57(2):80-9. doi: 10.1159/000077545. PMID 15192280
- [Background] Jiang Y, Wilk JB, Borecki I, Williamson S, DeStefano AL, Xu G, Liu J, Ellison RC, Province M, Myers RH. Common variants in the 5' region of the leptin gene are associated with body mass index in men from the National Heart, Lung, and Blood Institute Family Heart Study. Am J Hum Genet. 2004 Aug;75(2):220-30. doi: 10.1086/422699. Epub 2004 Jun 11. PMID 15197684
- [Background] Djousse L, Arnett DK, Eckfeldt JH, Province MA, Singer MR, Ellison RC. Alcohol consumption and metabolic syndrome: does the type of beverage matter? Obes Res. 2004 Sep;12(9):1375-85. doi: 10.1038/oby.2004.174. PMID 15483202
- [Background] Djousse L, Pankow JS, Arnett DK, Eckfeldt JH, Myers RH, Ellison RC. Apolipoprotein E polymorphism modifies the alcohol-HDL association observed in the National Heart, Lung, and Blood Institute Family Heart Study. Am J Clin Nutr. 2004 Dec;80(6):1639-44. doi: 10.1093/ajcn/80.6.1639. PMID 15585780
- [Background] Arnett DK, Miller MB, Coon H, Ellison RC, North KE, Province M, Leppert M, Eckfeldt JH. Genome-wide linkage analysis replicates susceptibility locus for fasting plasma triglycerides: NHLBI Family Heart Study. Hum Genet. 2004 Nov;115(6):468-74. doi: 10.1007/s00439-004-1182-y. Epub 2004 Sep 16. PMID 15375693
- [Background] Knox SS, Weidner G, Adelman A, Stoney CM, Ellison RC. Hostility and physiological risk in the National Heart, Lung, and Blood Institute Family Heart Study. Arch Intern Med. 2004 Dec 13-27;164(22):2442-8. doi: 10.1001/archinte.164.22.2442. PMID 15596634
- [Background] Djousse L, Arnett DK, Pankow JS, Hopkins PN, Province MA, Ellison RC. Dietary linolenic acid is associated with a lower prevalence of hypertension in the NHLBI Family Heart Study. Hypertension. 2005 Mar;45(3):368-73. doi: 10.1161/01.HYP.0000154679.41568.e6. Epub 2005 Jan 17. PMID 15655119
- [Background] Lin JP, Myers RH, Almasy L, Coon HH, Arnett DK, Hong Y, Hunt SC. Linkage of the cholesterol 7alpha-hydroxylase gene and low-density lipoprotein cholesterol conditional on apolipoprotein E association: the National Heart, Lung, and Blood Institute Family Heart Study. Chin Med J (Engl). 2005 Mar 5;118(5):362-9. PMID 15780204
- [Background] Djousse L, Rautaharju PM, Hopkins PN, Whitsel EA, Arnett DK, Eckfeldt JH, Province MA, Ellison RC; Investigators of the NHLBI Family Heart Study. Dietary linolenic acid and adjusted QT and JT intervals in the National Heart, Lung, and Blood Institute Family Heart study. J Am Coll Cardiol. 2005 May 17;45(10):1716-22. doi: 10.1016/j.jacc.2005.01.060. PMID 15893192
- [Background] Ellison RC, Zhang Y, Wagenknecht LE, Eckfeldt JH, Hopkins PN, Pankow JS, Djousse L, Carr JJ. Relation of the metabolic syndrome to calcified atherosclerotic plaque in the coronary arteries and aorta. Am J Cardiol. 2005 May 15;95(10):1180-6. doi: 10.1016/j.amjcard.2005.01.046. PMID 15877990
- [Background] Djousse L, Arnett DK, Carr JJ, Eckfeldt JH, Hopkins PN, Province MA, Ellison RC; Investigators of the NHLBI FHS. Dietary linolenic acid is inversely associated with calcified atherosclerotic plaque in the coronary arteries: the National Heart, Lung, and Blood Institute Family Heart Study. Circulation. 2005 Jun 7;111(22):2921-6. doi: 10.1161/CIRCULATIONAHA.104.489534. Epub 2005 May 31. PMID 15927976
- [Derived] Qavi AH, Zhou G, Ward RE, Carr JJ, Ellison RC, Arnett DK, Gaziano JM, Djousse L. Association of potato consumption with calcified atherosclerotic plaques in the coronary arteries: The NHLBI Family Heart Study. Nutr Metab Cardiovasc Dis. 2023 Dec;33(12):2413-2418. doi: 10.1016/j.numecd.2023.07.027. Epub 2023 Jul 25. PMID 37580232
- [Derived] Fretts AM, Follis JL, Nettleton JA, Lemaitre RN, Ngwa JS, Wojczynski MK, Kalafati IP, Varga TV, Frazier-Wood AC, Houston DK, Lahti J, Ericson U, van den Hooven EH, Mikkila V, Kiefte-de Jong JC, Mozaffarian D, Rice K, Renstrom F, North KE, McKeown NM, Feitosa MF, Kanoni S, Smith CE, Garcia ME, Tiainen AM, Sonestedt E, Manichaikul A, van Rooij FJ, Dimitriou M, Raitakari O, Pankow JS, Djousse L, Province MA, Hu FB, Lai CQ, Keller MF, Perala MM, Rotter JI, Hofman A, Graff M, Kahonen M, Mukamal K, Johansson I, Ordovas JM, Liu Y, Mannisto S, Uitterlinden AG, Deloukas P, Seppala I, Psaty BM, Cupples LA, Borecki IB, Franks PW, Arnett DK, Nalls MA, Eriksson JG, Orho-Melander M, Franco OH, Lehtimaki T, Dedoussis GV, Meigs JB, Siscovick DS. Consumption of meat is associated with higher fasting glucose and insulin concentrations regardless of glucose and insulin genetic risk scores: a meta-analysis of 50,345 Caucasians. Am J Clin Nutr. 2015 Nov;102(5):1266-78. doi: 10.3945/ajcn.114.101238. Epub 2015 Sep 9. PMID 26354543
- [Derived] Tanaka T, Ngwa JS, van Rooij FJ, Zillikens MC, Wojczynski MK, Frazier-Wood AC, Houston DK, Kanoni S, Lemaitre RN, Luan J, Mikkila V, Renstrom F, Sonestedt E, Zhao JH, Chu AY, Qi L, Chasman DI, de Oliveira Otto MC, Dhurandhar EJ, Feitosa MF, Johansson I, Khaw KT, Lohman KK, Manichaikul A, McKeown NM, Mozaffarian D, Singleton A, Stirrups K, Viikari J, Ye Z, Bandinelli S, Barroso I, Deloukas P, Forouhi NG, Hofman A, Liu Y, Lyytikainen LP, North KE, Dimitriou M, Hallmans G, Kahonen M, Langenberg C, Ordovas JM, Uitterlinden AG, Hu FB, Kalafati IP, Raitakari O, Franco OH, Johnson A, Emilsson V, Schrack JA, Semba RD, Siscovick DS, Arnett DK, Borecki IB, Franks PW, Kritchevsky SB, Lehtimaki T, Loos RJ, Orho-Melander M, Rotter JI, Wareham NJ, Witteman JC, Ferrucci L, Dedoussis G, Cupples LA, Nettleton JA. Genome-wide meta-analysis of observational studies shows common genetic variants associated with macronutrient intake. Am J Clin Nutr. 2013 Jun;97(6):1395-402. doi: 10.3945/ajcn.112.052183. Epub 2013 May 1. PMID 23636237